CLINICAL TRIAL: NCT03747276
Title: Can Electronic Information Kiosks Enhance Patient Accrual for Cancer Clinical Trials? A Pilot and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Information Kiosk
Record Dates: First submitted 2018-06-13; First posted 2018-11-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2018-11

CONDITIONS: Malignant Neoplasm
Keywords: clinical trial; accrual
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Trial Kiosk (Other)
  Interventions: Other: Clinical Trial Kiosk

INTERVENTIONS:
Other: Clinical Trial Kiosk — Kiosk will consist of a patient facilitator and a computer with access to general information about clinical trials and information specific to active clinical trials at the facility. Patients will be made aware of the kiosk via a large banner visible in the clinic above the kiosk.

SUMMARY:
The proposed study will include patients with non-haematologic cancer. Eligible patients will be invited to consent for participation in our study using standard demographic data collection forms and patient satisfaction questionnaires.

Cancer patients interested in learning more about clinical trials would be invited to go to the kiosk. A summer student approved and hired according to London Health Sciences Centre LHSC/Lawson criteria will be available from 0900-1630 daily for general assistance. If the student is overwhelmed by questions or numbers of patients, the Research Navigator or designate would be called to assist.

An information kiosk will be placed at the patient library on the ground floor of the LRCP. This kiosk will be outfitted with a computer and signage briefly outlining the title and purpose of the kiosk. Cancer patients interested in learning more about clinical trials would be invited to participate in our study by signing a consent form allowing the Research Navigator to contact them if they expressed interest in knowing more about a clinical trial.

DETAILED DESCRIPTION:
The proposed study will include patients with non-haematologic cancer. Eligible patients will be invited to consent for participation in our study using standard demographic data collection forms and patient satisfaction questionnaires.

Cancer disease site teams (DSTs) were asked to prioritize trials that open from May 1 to Sept.30, 2018 and likely to accrue three patients over six months for major accruing tumour sites (lung, breast, GI, GU, melanoma and symptom control/supportive care/multi-site such as oligometastatic) and one patient over six months for other sites.

Patients are made aware of the kiosk via advertising in the facility including a card given at registration each day outlining the existence, location and purpose of the kiosk. The location will be marked by visual cues (banner and balloons). Cancer patients interested in learning more about clinical trials would be invited to go to the kiosk. A summer student approved and hired according to LHSC/Lawson criteria will be available from 0900-1630 daily from July 3-Aug 31 for general assistance. If the student is overwhelmed by questions or numbers of patients, the Research Navigator or designate would be called to assist.

An information kiosk will be placed at the patient library on the ground floor of the LRCP. This kiosk will be outfitted with a computer and signage briefly outlining the title and purpose of the kiosk. Cancer patients interested in learning more about clinical trials would be invited to participate in our study by signing a consent form allowing the Research Navigator to contact them if they expressed interest in knowing more about a clinical trial. They would still be able to read a lay online or printed paper document giving them background information on clinical trials (i.e. what is a clinical trial?) whether they consented or not. To save on resources, the pilot will utilize general information available to the public from the Stanford Cancer Institute Clinical Trials website at http://med.stanford.edu/cancer/trials.html and a Canadian website http://itstartswithme.ca/why-participate/ . Information specific to clinical trials at London Regional Cancer Program (LRCP) will be made available by linking to an internal resource. Patients will be asked if they would be interested in seeing brief summaries of selected clinical trials currently available at the LRCP. They would then be asked to review a list of possible trials they may be eligible for based on their cancer diagnosis. Patients will have the option to click on each of the applicable trials to obtain more information including: trial title, NCT number, a lay description, why the study is important, principal investigator name, and a short list of eligibility criteria. Additionally, patients have the option to send any trial information they might be interested in to their home their email address or obtain a paper copy of the information.

Finally, at the kiosk patients who signed a consent, would have the option to submit electronically their first/last name and DOB in order to grant permission for a member of the Clinical Research Unit (CRU) staff, the Research Navigator, to review their request for further clinical trial information, contact them with potential options and contact their oncologist(s) to discuss their potential enrollment in a specific trial. This consent, patient name and PIN numbers would then be emailed to the CRU. Alternatively, they could fill this out on a paper form that would be dropped into a secure mailbox at the kiosk that would be collected at the end of each day. The information would be logged on a secure electronic database by HM and the paper documents except for consent destroyed (or kept in a secure area). The Research Navigator would contact the patient by phone to provide further details of the trial(s) of interest and to determine eligibility. If the patient is interested and eligible, an indication of the clinical trial of interest would be added to the scheduling list beside the patient's name.

After a two week run in phase, accrual, logistical and communications issues will be reviewed to ensure the kiosk project is functioning efficiently and to review patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with a solid tumour cancer (including breast, central nervous system, gynecologic, gastrointestinal, genitourinary, head and neck, liver, melanoma, neuroendocrine, sarcoma, thoracic, thyroid).
* Patients able to provide independent informed consent.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients diagnosed with haematologic malignancy unless there is a co-existing solid tumour cancer
* Inability to provide informed consent
* Inability to read and comprehend written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-11-18 (Actual)

PRIMARY OUTCOMES:
Change in accrual rate | 4 months (A two month rate of accrual (May-June, 2018) will be determined before opening the kiosk. A second two month accrual period (August-September) will be used to assess the change in trial accrual.
  Our primary objective is to quantify the clinical trial accrual rates in a subset of trials that are selected as priority trials and are open both two months before and three months after implementation of the clinical trial information kiosk. Accrual rates before and after implementation will be compared.

SECONDARY OUTCOMES:
Proportion of patients requesting research navigator contact | 3 months
  1. To determine the proportion of patients who accessed the kiosk provided information so that they could be contacted by the Research Navigator.
Proportion of patients contacted eligible for clinical trial | 3 months
  2. To determine what proportion of patients who were contacted the research navigator were eligible to participate in a clinical trial.
Proportion of eligible patients participating in clinical trial | 5 months
  To determine what proportion of patients eligible for a clinical trial actually participated.
Satisfaction with kiosk | 2 months
  To evaluate patient satisfaction with the clinical trial information kiosk using a Likert scale.
Proportion of patients accessing kiosk | 2 months
  To determine the number of individuals who interacted with the information kiosk compared to total number of cancer patients seen in clinic when the kiosk is open.

OTHER OUTCOMES:
Demographics | 2 months
  Demographic correlations of patients seeking additional information. This will include age, sex, urban/rural status obtained from electronic health records. Patients will also be asked to voluntarily provide information on income, occupational status and whether they had previously been approached about a cancer clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Present at meetings and publish in peer reviewed journal
Supporting Information: Study Protocol
Time Frame: One year